CLINICAL TRIAL: NCT06794216
Title: Comparison of Expanded Hemodialysis With 3 Other Dialysis Techniques in the Removal of Uremic Toxins in Chronic Renal Failure
Brief Title: Comparison of Hemodialysis Techniques in the Removal of Uremic Toxins in Chronic Renal Failure
Acronym: EMPIRE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EMPIRE
Record Dates: First submitted 2024-12-30; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, expanded hemodialysis has been the subject of studies, many of them done on small populations, with limited observation periods and not always unambiguous results. In the literature, there are data comparing HDx and high-flow hemodialysis in terms of small- and medium-molecule purification and control of inflammation indices; there are fewer data comparing HDx and HDF online. In contrast, there are no studies in the literature comparing HDx with HFR. With a view to personalizing therapy, demonstrating the equivalence/superiority of HDx over the other dialysis techniques under consideration could make this technique suitable precisely for that class of more malnourished and more frail patients who to date do not obtain benefits from the other methods.

The objective of the study is the mid-term (12-month) evaluation and comparison of the MCO filter called Theranova 400™ (1.7 m2, steam sterilization, cut-off 25 Kda, Baxter, Heichingen, Germany) with high-flux hemodialysis (HF-HD), OL- HDF and hemodiafiltration with endogenous reinfusion (HFR) with HFR filter 17 , in combination with medical therapy under normal clinical practice, in terms of purification of low and medium molecular weight uremic toxins, control of baseline inflammatory status and erythropoietin resistance in patients with chronic renal failure undergoing hemodialysis treatment.

DETAILED DESCRIPTION:
Data from approximately 50 patients with chronic end-stage renal disease treated consecutively during the considered study period with HDx with Theranova filter, with HF HD, with OL-HDF, and with HFR with HFR17 filter at the Dialysis Center of the O.U. of Nephrology, Dialysis and Transplantation, directed by Prof. Gaetano La Manna, of IRCCS AOUBO Policlinico Sant'Orsola in the period from 01/01/2018 to 30/11/2022 will be analyzed. It should be noted that these membranes were used as part of the normal course of care.

The study is observational, non-interventional in nature. Patients will be treated according to clinical practice in accordance with the judgment of the physician and the information in the Technical Data Sheet of each individual product of any concomitant therapies administered according to clinical practice.

There will be about 50 patients, divided into 4 cohorts: patients undergoing HDx treatment with Theranova filter (group A), patients undergoing HFR treatment with HFR17 filter (group B), patients undergoing OL- HDF treatment (group C) and patients undergoing HD treatment with HF filter (HF HD) (group D). Each group will consist of at least 10 patients with chronic terminal kidney disease undergoing dialysis treatment at the O.U. of Nephrology, Dialysis and Transplantation, directed by Prof. Gaetano La Manna, of IRCCS AOUBO Policlinico Sant'Orsola from 01/01/2018 to 30/11/2022.

Inclusion criteria.

* Age ≥ 18 years
* Chronic hemodialytic treatment (on dialysis for at least 6 months), hemodialytic treatment with MCO filter (Theranova) or HF filter, OL- HDF or HFR with HFR filter17.
* Continuous use of the same filter for at least 12 months.
* Diuresis < 200 ml/day.
* Tri-weekly hemodialysis treatment.
* Duration of session ≥ 210 minutes.
* Availability of clinical data collected during the follow-up occurred at the OU of Nephrology, Dialysis and Transplantation - La Manna.

Exclusion criteria.

* Intradialytic hypotension
* Need for dialysis without heparin
* Active bleeding
* Active hematologic diseases
* Thrombocytopenia
* Chronic hepatopathies
* Active systemic inflammatory diseases
* Uncontrolled diabetes mellitus
* Temporary vascular access
* Recurrent vascular access infections

A sample size of approximately 50 patients treated consecutively during the study period under consideration and within the inclusion criteria with HDx with Theranova filter, HF HD, OL-HDF or HFR with HFR filter17 is estimated. The study will be initiated after formal notification to the Ethics Committee. Only patients undergoing chronic dialysis treatment at the OU of Nephrology, Dialysis and Transplantation, directed by Prof. Gaetano La Manna, of IRCCS AOUBO Policlinico Sant'Orsola will be enrolled.

Study Duration:

Patient data will be collected for the period from 01/01/2018 to 30/11/2022. A total duration of 18 months is estimated for data collection and analysis, starting from the approval of the Ethics Committee and issuance of the Nulla Osta by the General Management.

Treatments, visits and evaluations:

There are no study-specific treatments other than those provided by normal clinical practice.

For the purpose of this clinical trial, no study-specific visits are planned, but patients eligible in the study, still in follow-up, will be asked to read the information sheet and sign a study-specific informed consent for the collection and evaluation of the specified clinical-anamnestic data specified below. Clinical data will be collected in a structured manner from patients' medical records. It is specified that patient data will be collected for the period from 01/01/2018 to 30/11/2022.

The clinical data required by the protocol will be collected in pseudonymized form by the Principal Investigator's designated personnel in an electronic Data Collection Form (CRF) and will be managed through the REDCap platform. The eCRF in REDCap will be requested and implemented according to the procedure described in the "Corporate Operational Instruction for the Management and Use of the REDCap Platform" (IOA119). The Principal Investigator must indicate the names of personnel delegated to data management by specifying their relative functions within the study in the Delegation log.

Analysis Methodology:

The demographic and clinical characteristics of patients treated in the period 01/01/2018- 30/11/2022 at the Center, enrolled and evaluated in the study, will be reported in summary tables. Given the large number of patients under study (n=10 per group), descriptive statistics such as median, minimum value and maximum value for continuous type variables; absolute frequencies and percentage relative frequencies (when appropriate) for discrete or nominal type variables will be reported.

Summary data of blood parameters, relevant clinical events, etc., taken during the observation period will be summarized in summary tables.

Summary data of blood parameters, relevant clinical events, etc., collected during the observation period will be summarized in summary tables.

Data analysis will be carried out using SPSS software. For variables with normal distribution the Anova test will be used, for variables with distribution the Kruskal-Wallis test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Chronic hemodialytic treatment (on dialysis for at least 6 months), hemodialytic treatment with MCO filter (Theranova) or HF filter, OL- HDF or HFR with HFR filter17.
* Continuous use of the same filter for at least 12 months.
* Diuresis < 200 ml/day.
* Trisweekly hemodialysis treatment.
* Session duration ≥ 210 minutes.
* Availability of clinical data collected during the follow-up that took place at the O.U. of Nephrology, Dialysis and Transplantation - La Manna

Exclusion Criteria:

* Intradialytic hypotension
* Need for dialysis without heparin
* Active bleeding
* Active hematologic diseases
* Thrombocytopenia
* Chronic hepatopathies
* Active systemic inflammatory diseases
* Uncontrolled diabetes mellitus
* Temporary vascular access
* Recurrent vascular access infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be about 50 patients, divided into 4 cohorts: patients undergoing HDx treatment with Theranova filter (group A), patients undergoing HFR treatment with HFR17 filter (group B), patients undergoing OL- HDF treatment (group C) and patients undergoing HD treatment with HF filter (HF HD) (group D). Each group will consist of at least 10 patients with chronic terminal kidney disease undergoing dialysis treatment at the O.U. of Nephrology, Dialysis and Transplantation, directed by Prof. Gaetano La Manna, of IRCCS AOUBO Policlinico Sant'Orsola from 01/01/2018 to 30/11/2022.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference between Dialysis' methods | Baseline (0 months), 3 months and 12 months
  For the blood parameters of interest, taken at pre-dialysis and over the long interdialytic period at the end of dialysis during follow-up, changes will be analyzed by Wilcoxon tests (e.g., pre-dialysis uremic toxins with blood levels of the same substances at the end of dialysis or with their respective RRs) to assess the magnitude of differences found before and after dialysis. A comparison will be made between patients treated with the same dialysis technique and then a comparison with patients treated with the other methods examined considering time 0 and then at 3 and 12 months after the start of treatment with the same filter and dialysis method. The percentage of change in the medium term of erythropoietin dose and ev administered iron, the change in ERI and martial balance will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano La Manna, MD, Principal Investigator — IRCCS AOU di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Emilia-Romagna, Italy